CLINICAL TRIAL: NCT04286087
Title: Assessment of Clinical Outcomes in Closure of Deep Neck Space Infection Incisions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Dr Rudecki, the principal PI has left the program and is no longer in the United States therefore he failed to recruit patients for the study.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Craig Bradley Pearl, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-DB-19-1029
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Deep Neck Space Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Arm (Experimental)
  Interventions: Procedure: neck incisions closed at bedside at the time of drain removal under local anesthesia
- Control Group (Active Comparator)
  Interventions: Procedure: standard treatment

INTERVENTIONS:
Procedure: neck incisions closed at bedside at the time of drain removal under local anesthesia — Participants allocated to the investigational group will have neck incisions closed at bedside at the time of drain removal under local anesthesia
  Arms: Investigational Arm
Procedure: standard treatment — Participants in the control group will have standard treatment performed as per current practice,their incision will be left to close by secondary intention
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine if closure of deep neck infection incisions at the time of extraoral drain removal has any impact on rates of reinfection and to determine if this treatment will have any impact on scar formation and qualitative measures of pain or impact on quality of life during the post-operative healing period.

ELIGIBILITY:
Inclusion Criteria:

* deep neck space infection
* who require a conservative unilateral submandibular neck incision to access affected deep fascial neck spaces

Exclusion Criteria:

* pregnant females
* cognitively impaired individuals
* deep neck space infections which require bilateral neck incisions, large neck apron incisions, or placement of negative pressure therapy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-09 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with reinfection | 1-2 weeks post intervention

SECONDARY OUTCOMES:
Number of participants requiring a scar revision surgery | 4-6 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Craig Pearl, BDS, Principal Investigator — The University of Texas Health Science Center, Houston

IPD SHARING:
Plan to Share IPD: No